CLINICAL TRIAL: NCT07327008
Title: Investigation of the Effectiveness of the Telerehabilitation Program in Patients With Liver Transplantation
Brief Title: The Effectiveness of Telerehabilitation in Liver Transplant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Alper AYAS, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-AA-01
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation; Telerehabilitation
Keywords: liver transplantation; telerehabilitation; exercise; quality of life
MeSH Terms: conditions — Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: There are two groups: a telerehabilitation group and home exercise program group.
Who Masked: Outcomes Assessor
Masking Description: Our study has two groups. The results will be evaluated by a blinded researcher who does not know which group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): The telerehabilitation group will receive videoconference-based telerehabilitation three days a week for eight weeks. All exercises will be performed under the supervision of a physiotherapist.
  Interventions: Other: Telerehabilitation
- Home exercise program group (Active Comparator): Home exercise program group will initially be given instructions on the exercises and asked to perform them three days a week for eight weeks. They will be contacted by phone once a week to inquire whether they are doing the exercises.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Telerehabilitation — The telerehabilitation program will include breathing, strengthening, balance, and walking exercises, with increasing intensity week by week, and stretching exercises targeting major muscles will be given during the cool-down period.
  Arms: Telerehabilitation group
Other: Home exercise — Patients will be given brochures on breathing, strengthening, balance and walking exercises and asked to perform them without a physiotherapist.
  Arms: Home exercise program group

SUMMARY:
Liver transplantation is defined as a surgical procedure in which a liver with tissue damage and inability to perform its functions is replaced, in whole or in part, with a healthy liver obtained from a living or deceased donor. Post-transplantation treatment includes medical treatment, physiotherapy, and rehabilitation. Physiotherapy and rehabilitation, an important component of liver transplantation management, consists of three phases: preoperative, early postoperative, and late postoperative. Telerehabilitation is currently defined as the control or monitoring of rehabilitation remotely using telecommunication-related technologies. Studies on telerehabilitation in liver transplant patients are insufficient in the literature. The aim of this study is to investigate the effect of a telerehabilitation-based exercise program applied to liver transplant patients on exercise capacity, respiratory muscle strength, peripheral muscle strength, fatigue level and quality of life.

DETAILED DESCRIPTION:
Participants will be randomly divided into two groups: a telerehabilitation group and home exercise program group. Both groups will be evaluated before and after treatment (week 8). The telerehabilitation group will receive videoconference-based telerehabilitation three days a week for eight weeks. All exercises will be performed under the supervision of a physiotherapist. Each telerehabilitation session will last approximately 30-45 minutes. The exercises will be performed in the following order: breathing exercises, strengthening exercises, balance exercises, and walking exercises. The home exercise program group will receive an exercise brochure after the initial evaluation. Both groups will continue with their standard medical treatments, and a second evaluation will be conducted at the end of eight weeks. Participants' exercise capacity will be assessed using the "6-Minute Walk Test," fatigue level using "The Fatigue Severity Scale", respiratory muscle strength by measuring "Maximal inspiratory pressure (MIP)" and "Maximal expiratory pressure (MEP)", muscle strength using a digital dynamometer, balance using the "Timed Up and Go Test," and quality of life using the "The Liver Disease Symptom Index 2.0"

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age and having undergone a liver transplant
* Having had a liver transplant operation at least 6 months prior
* Spontaneous breathing
* Hemodynamic stability
* Reading and writing skills
* Ability to mobilize independently, ability to follow verbal and visual instructions

Exclusion Criteria:

* Presence of unstable cardiovascular disease
* Presence of primary lung disease requiring regular bronchodilator treatment
* Presence of neuromuscular disease or neurological complications
* Musculoskeletal limitation/use of assistive devices
* Being a multiple organ transplant recipient
* Presence of orthopedic disability and functional capacity limitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | eight weeks
  Exercise capacity will be assessed using the Six-Minute Walk Test, which plays an important role in evaluating pre- and post-operative exercise performance in liver transplant patients. The test will be conducted in a 30 m long, enclosed, straight corridor under the supervision of a physiotherapist, in accordance with the criteria set by the American Thoracic Society. The patients' heart rate and peripheral capillary oxygen saturation values will be recorded before, during, and after the test using a portable pulse oximeter. Dyspnea and perceived fatigue levels will be assessed using the Modified Borg Scale (MBS) during the test. The total walking distance completed in six minutes will be recorded in meters as the individual's six-minute walk distance
Timed Up and Go Test | eight weeks
  Used to evaluate the balance performance of individuals during movement. The person sits in a chair of standard height (46 cm), a distance of 3 meters is measured from the chair and a cone is placed at the end of this distance to indicate it. After receiving the command "walk as fast as you can and sit back down in the chair," the person gets up, walks down the corridor for meters, turns around, walks back to the chair and sits down. The time from the moment of getting up from the chair until the person turns around and sits back down in the chair is measured with a stopwatch and recorded in seconds.

SECONDARY OUTCOMES:
The Liver Disease Symptom Index 2.0 | eight weeks
  The Chronic Liver Disease Quality of Life Scale 2.0 will be used as a disease-specific measurement tool. It is a scale developed to objectively evaluate the clinical and psychological consequences on physical and daily living activities in chronic liver disease and to determine the severity of the disease. The Chronic Liver Disease Quality of Life Scale 2.0 , which has been applied in different stages of chronic liver diseases and psychometrically tested, evaluates the effects of symptoms on daily life as well as symptom severity. It is a useful and practical scale in clinical use, whose validity and reliability have been established in the Turkish population
The Fatigue Severity Scale | eight weeks
  The Fatigue Severity Scale (FSS) is a nine-item self-administered scale. The scale correlates moderately well with the Visual Analog Scale (VAS) and is therefore a good tool for assessing the severity of fatigue. Patients are asked to choose a number from 1 to 7 indicating how much they agree or disagree with the statement. "1 point" indicates strong disagreement, "7 points" indicates strong agreement. A score of 4 and above generally indicates severe fatigue.
Respiratory Muscle Strength Measurement | eight weeks
  Respiratory muscle strength will be assessed by measuring the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), which are intraoral pressure measurements. The measurement will be performed using a portable intraoral pressure gauge with the maximal breathing method while the airway is closed with a valve.
Muscle Strength Measurement | eight weeks
  This is a method used to measure muscle strength in patients. A La Fayette handheld digital dynamometer will be used during the test. To obtain isometric contraction during the test, the person performing the measurement is asked to hold the dynamometer steady while the person being tested applies maximum contraction against the device. The patient will be asked to hold the maximal isometric contraction for 5 seconds, followed by a 30-second rest interval and the same procedure will be repeated 3 times on the dominant side and the average of the measurement values will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Faculty of Health Sciences, Physiotherapy and Rehabilitation Laboratory, Büyükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No